CLINICAL TRIAL: NCT07367308
Title: The Effect of External and Combined Focus Instructions on Lower Extremity and Trunk Kinetic and Kinematic Parameters During Landing in Young Female Athletes With Asymptomatic Dynamic Knee Valgus - A Randomized Controlled Trial
Brief Title: External vs Combined Focus Effects on Landing in Female Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: California State University, Long Beach (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSCSULB-2026
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Valgus Deformity, Not Elsewhere Classified, Knee; Injury, Knee
Keywords: cue; Motor Learning; skill transfer
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Female athletes meeting the inclusion criteria will be randomized into the combined attentional focus group, the external attentional focus group, and the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Focus of Attention Group (CFAG) (Experimental): After participants meet the inclusion criteria are randomized and assigned to the combined attentional focus group. They will perform training blocks consisting of 5 repetitions and 2 sets of single-leg drop jump landings before and after the evaluations. During the jumps, instructions will focus on combined attentional focus and will be repeated for each jump. A 1-minute rest period will be provided between training blocks.
  Interventions: Other: Single-Leg Drop Vertical Jump; Other: Combined Focus of Attention Instruction
- External Focus o Attention Group (EFAG) (Experimental): After participants meet the inclusion criteria are randomized and assigned to the external attentional focus group. They will perform training blocks consisting of 5 repetitions and 2 sets of single-leg drop jump landings before and after the evaluations. During the jumps, instructions will focus on external attentional focus and will be repeated for each jump. A 1-minute rest period will be provided between training blocks.
  Interventions: Other: Single-Leg Drop Vertical Jump; Other: External Focus of Attention Instruction
- Control Group (Active Comparator): After participants meet the inclusion criteria are randomized and assigned to the control group. They will perform training blocks consisting of 5 repetitions and 2 sets of single-leg drop jump landings before and after the intervention. During the jumps, no instructions will be given. A 1-minute rest period will be provided between training blocks.
  Interventions: Other: Single-Leg Drop Vertical Jump; Other: No instruction

INTERVENTIONS:
Other: Single-Leg Drop Vertical Jump — Single-Leg Drop Vertical Jump test will be performed with the dynamic knee valgus leg.
Other: Combined Focus of Attention Instruction — - Combined focus group: "When you land, keep your knee over your toes while directing your knee toward the cone."
  Arms: Combined Focus of Attention Group (CFAG)
Other: External Focus of Attention Instruction — - External focus group: "When you land, direct your movement toward the cone placed on your side."
  Arms: External Focus o Attention Group (EFAG)
Other: No instruction — Control group: No specific instructions.
  Arms: Control Group

SUMMARY:
Female athletes are at higher risk of knee injuries, particularly non-contact anterior cruciate ligament (ACL) injuries, often caused by dynamic knee valgus during landing. Proper landing techniques and neuromuscular training are crucial for injury prevention. Attentional focus strategies, such as external focus (EF) and internal focus (IF), can influence movement patterns, muscle activation, and skill transfer during landing tasks. EF generally promotes safer and more controlled landings, while IF offers certain kinematic benefits. However, real-world sports often require a combination of attentional strategies, and the effects of combined EF + IF instructions on landing mechanics and muscle activation have not been fully studied.

This study will investigate the effects of EF and combined attentional focus instructions on lower extremity and trunk movement, muscle activation, and skill transfer in young female athletes with asymptomatic dynamic knee valgus. The investigators aim to determine whether combined attentional focus training provides greater improvements in landing mechanics, muscle activation, and skill transfer than EF training alone.

DETAILED DESCRIPTION:
Female athletes experience knee injuries significantly more often, with an incidence rate approximately 3.5 times higher than that of their male counterparts. One of the most common knee injuries is anterior cruciate ligament (ACL) injury, with the risk being particularly high in female athletes, who have a reported incidence of non-contact ACL injuries of 63%.

Approximately 70% of ACL injuries occur without contact, with one of the most frequent causes being dynamic knee valgus which can result in high abduction (valgus) loads during landing after a jump. Dynamic knee valgus describes the frontal-plane knee angle during dynamic tasks such as landing or stepping down, typically occurring in conjunction with femoral internal rotation, contralateral pelvic drop, and hip adduction. Female athletes exhibit significantly greater valgus angles than male athletes, with only 22% of female players classified as having good knee control during jump landing, compared with 80% of male players.

The initial landing phase after a jump requires special attention from injury-prevention professionals, as 31% of ACL injuries occur during this phase. Common biomechanical features during single-leg landing include decreased flexion angles of the ankle, knee, hip, and trunk; increased knee internal rotation and abduction (valgus) angles and moments; lateral trunk flexion; as well as exaggerated ground reaction forces. An important clinical implication of these findings is that athletes need to be taught safer landing techniques.

Recently, the importance of integrating cognitive strategies into injury prevention programs has been emphasized. One such cognitive strategy involves the external and internal focus of attention, in which instructions for executing the movement aim to improve neuromuscular performance and motor learning. In external focus (EF), the athlete's attention is directed to objects or the environment external to the body (e.g., "stand on one leg and slowly bend your knee while keeping your knee over your foot"), while in internal focus (IF), attention is directed toward the performer's own movements (e.g., "stand on one leg and reach slowly toward the cone with your knee while bending your knee").

Previous studies reported that EF and IF instructions have different effects on athletes' kinematic, kinetic, and muscle activation parameters. EF instructions enhance safer and more controlled movement patterns during jump-landing by increasing knee and hip flexion, reducing knee valgus moments, and increasing the overall range of motion compared to IF. IF instructions, on the other hand, may provide certain kinematic improvements, such as reducing knee varus moments and controlling medial-lateral displacement. Recent meta-analyses support these findings, showing that although EF is generally more effective in jumping tasks, both attentional focus types can improve knee flexion.

However, real-world sports environments are complex, requiring athletes to dynamically shift attention between IF and EF or use both simultaneously. Evidence supports the effectiveness of dynamic attentional use and highlights the need for further research investigating combined attentional focus strategies. The acute and one-week effects of combined attentional focus and video-based instructions, finding that verbal combined focus instructions produced greater improvements in DK and landing performance. Since female athletes demonstrated higher incidence rate of ACL injury and more commonly present with dynamic knee valgus, there is a need for sex-specific studies investigating the effects of combined attentional focus training on kinetic and kinematic parameters in individuals with dynamic knee valgus.

Previous studies also reported that EF and IF instructions result in difference muscle activation. It is reported that EF not only increases knee and hip flexion but also enhances the feedforward activation of the gluteus medius and gluteus maximus muscles, resulting in safer and more controlled landing mechanics. Although IF provides certain kinematic improvements and can enhance quadriceps activation in isokinetic settings, its effects on EMG activation are less pronounced than those observed with EF. Therefore, EF seems to offer clearer advantages in terms of both motor efficiency and muscle activation. However, to our knowledge, no study has examined the effects of combined attentional focus instructions on muscle activation outcomes, highlighting an important area for future research.

Skill transfer, or the ability to generalize learned motor patterns to new or more complex tasks, is a critical indicator of effective motor learning and real-world performance. Improvements in jump-landing technique successfully transferred to a sidestep cutting task when athletes were trained with EF or video-based instructions, suggesting that EF facilitates safer and more efficient motor performance in dynamic conditions. More research is needed to determine how skill acquisition interventions can optimize the generalization of learned motor skills and to understand the influence of combined attentional focus instructions on skill transfer outcomes.

In this study, The investigators aimed to investigate the effects of EF and combined attentional focus (EF + IF) instructions on lower extremity and trunk kinetic, kinematic, muscle activation parameters and skill transfer ability in young asymptomatic female athletes with dynamic knee valgus. The investigators hypothesized that combined attentional focus training would yield greater improvements in dynamic knee valgus and other associated biomechanical parameters, muscle activation and skill transfer than external focus training.

ELIGIBILITY:
Inclusion Criteria:

Females aged between 18-30 years old

BMI between 18.5-25 kg/m²

Dynamic knee valgus >10° during single-leg squat test (Richardson et al., 2020)

Being recreationally active (engage in moderate physical activities at least 3 times a week, with each session lasting at least 30 minutes in the past 4 weeks) (Heinert, 2008)

Exclusion Criteria:

Trunk, lower back, or lower extremity pain greater than 3/10 on numeric pain rating scale (0-10) in the past 6 months

History of surgeries in the lower extremity or lower back that may affect the landing mechanism

Currently participating in any lower extremity biomechanics modification program

Any medical or physical condition that would prevent safe jumping from a 20-cm box

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
3D motion analyses | baseline, immediately after the intervention, one week after the baseline
  3D motion analysis will be used to evaluate lower extremity and trunk kinematics and kinetics during a single-leg drop vertical jump task. Retroreflective markers will be placed on anatomical landmarks of the foot, shank, thigh, pelvis, trunk, upper extremity, and head using a standardized whole-body marker set. Marker trajectories will be captured using a multi-camera motion capture system synchronized with force platforms to record ground reaction forces. Following a static calibration trial, participants will perform three trials of a single-leg drop vertical jump from a 20-cm platform using the limb demonstrating dynamic knee valgus. Kinematic variables will include peak joint angles of the hip, knee, and ankle in sagittal, frontal, and transverse planes, as well as trunk motion. Kinetic variables will include hip and knee joint moments and peak vertical ground reaction force. Outcome measures will be averaged across trials for pre-, post-, and retention assessments.

SECONDARY OUTCOMES:
Gluteal muscle activation (EMG) | baseline, immediately after the intervention, one week after the baseline
  Surface electromyography (EMG) will be used to assess muscle activation of the gluteus medius and gluteus maximus during testing. EMG signals will be collected using a wireless multi-channel system. Prior to electrode placement, skin preparation will be performed to reduce impedance. Bipolar surface electrodes will be placed parallel to muscle fibers using standardized placement procedures, and correct positioning will be verified through voluntary muscle activation.
  Maximal voluntary isometric contractions (MVICs) will be performed for each muscle to normalize EMG data. Three MVIC trials of 5 seconds will be recorded with adequate rest between trials. EMG data will be synchronized with motion capture and force platform data. Muscle activation outcomes will be averaged across trials for pre-, post-, and retention assessments and used for subsequent analysis.
Forward Step-Down Test | baseline, immediately after the intervention, one week after the baseline
  Participants will stand on an 8-inch (20-cm) step with their hands placed on their hips. They will be instructed to lower the non-test leg until the heel lightly touches the floor and then return to the starting position, keeping the test leg on the step throughout the movement. A metronome will be used to standardize the movement speed, set at 60 beats per minute (1 second for descent and 1 second for ascent). The movement will be simultaneously recorded using a three-dimensional motion capture system (Qualisys, Gothenburg, Sweden) to collect kinematic data for the hip, knee, and ankle joints during the task.

OTHER OUTCOMES:
manipulation check | baseline, immediately after the intervention, one week after the baseline
  At the end of each training block and after the post-evaluation, participants' focus during the jumps will be assessed. All participants will be asked to indicate where they directed their attention during the jump. For the external focus group, options will be "cone" or "other (please specify)." For the combined focus group, options will be "cone," "knee," or "other (please specify)." The control group will also be asked to report where their attention was focused. In addition, participants in the external and combined focus groups will rate how closely they followed the instructions on a 0-10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PT, PhD, Principal Investigator — Bahçeşehir University; Sharon Teng, PT, PhD, Study Chair — California State University, Department of Physical Therapy
Locations (1):
- California State University, Long Beach, Long Beach, California, United States